CLINICAL TRIAL: NCT04121338
Title: Prospective Single-Arm Pilot Study for CT-Guided, Temporary Celiac Ganglion Block as a Test Before Celiac Ganglion Resection for Dysautonomia-Related Bowel Dysmotility
Brief Title: Temporary Celiac Ganglion Block as a Test Before Celiac Ganglion Resection for Dysautonomia-Related Bowel Dysmotility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00198738
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Dysautonomia
Keywords: celiac ganglion block; resection; bowel dysmotility
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: 10 patients with chronic GI dysmotility, chronic nausea/vomiting and feeding intolerance requiring G-J feeding and considered for Celiac Ganglion resection
Masking Description: Since this is a single arm study, no masking will be performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Test group (Experimental): 10 patients with presumptive diagnosis of dysautonomia with chronic nausea, vomiting and food intolerance
  Interventions: Procedure: Celiac ganglion block; Drug: Liposomal bupivacaine

INTERVENTIONS:
Procedure: Celiac ganglion block — The celiac ganglion block will be performed under CT guidance and with the patent under moderate sedation. With the patient prone the back will be prepped and draped sterility. Under CT guidance two 22 gauge needles will be placed with the tips on either side of the celiac artery. This is the location of the celiac ganglia. Liposomal bupivacaine will then be injected in that location. Maximum dose is 133 mg for 75 kg person. For lower weight patients, dose will be weight based. Then patient will be observed for 1-2 hours post procedure and then discharged to home
Drug: Liposomal bupivacaine — Liposomal bupivacaine will then be injected in that location. Maximum dose is 133 mg for 75 kg person. For lower weight patients, dose will be weight based.
  Other Names: Exparel

SUMMARY:
Dysautonomia is malfunction of the autonomic nervous system. It usually results from overactivity of the sympathetic portion and over-secretion of acetylcholine. Symptoms depend on the organ involved by this sympathetic overstimulation. Involvement of the gastrointestinal system results in chronic dysmotility, nausea, vomiting, food intolerance, weight loss and need for feeding tube placement and/or parenteral feeding. Autonomic celiac ganglia resection has been shown to alleviate symptoms as it interrupts the sympathetic stimulation to the gastrointestinal (GI) system, however there is no pre surgery test to confirm the diagnosis. The investigators' objective is to temporarily block the celiac ganglion with a long acting anesthetic (liposomal bupivacaine). If symptoms abate the diagnosis is confirmed and patient will proceed to surgery.

DETAILED DESCRIPTION:
Problem:

Dysautonomia is malfunction of the autonomic nervous system. It usually results from overactivity of the sympathetic portion and over-secretion of acetylcholine. Symptoms depend on the organ involved by this sympathetic overstimulation. A partial list of dysautonomia-related conditions is shown below:

Affected Level Manifestation Cardiac innervation Postural Orthostatic Tachycardia Syndrome Skin Hyperhidrosis Arteries Raynaud's phenomenon Kidneys Hypertension Small nerve fibers Reflex Sympathetic Dystrophy Pain fibers Complex regional pain syndrome GI system Chronic GI dysmotility/irritable bowel syndrome (IBS) The last one (Chronic GI dysmotility) usually affects young females, presenting after puberty. Symptoms include chronic abdominal pain, intestinal angina, chronic nausea/vomiting, inability to take po, need for total parenteral nutrition (TPN) or G-tube feeding. Further, the patients' condition is often complicated by opioid dependence, malnutrition, weight loss, social isolation etc. Many such patients are misdiagnosed as having Median Arcuate Ligament Syndrome (MALS) and are referred to surgery for ligament release. Though some of the patients do get partial relief, this temporary relief is due to the partial interruption of the sympathetic nerves during surgery. Repeat surgery to complete celiac ganglion resection is often necessary. Occasionally surgeons refer patients for a Computer Tomography (CT) guided temporary celiac ganglion block to confirm (or exclude) sympathetic system dysfunction as the cause of the patients symptoms. However negative or positive predictive value of this test has not been studies rigorously.

Research Hypothesis:

The investigators' hypothesis is that a low-risk, outpatient test can confirm (or exclude) dysautonomia as the cause of the patient's symptoms. The experimental test is CT-guided, celiac ganglion temporary block with liposomal bupivacaine.

Importance of the Research:

Some of the patients who are diagnosed as having MALS have in fact dysautonomia and have the wrong surgery. Many other patients with dysautonomia-related GI symptoms are not diagnosed at all and offered only symptomatic treatment. The development of CT-guided, celiac ganglion temporary block with liposomal bupivacaine as a low-risk confirmatory test for dysautonomia-related GI symptoms, will improve surgical outcomes and afford a novel treatment option to many patients.

2. Objectives

CT-guided, celiac ganglion temporary block with liposomal bupivacaine will eliminate sympathetic input to the bowel. Its half-life is 24 hours and therefore symptom relief can be distinguished from overlap due to procedural sedation.

Primary:

1. Improved tolerance to per os (PO) solid food intake
2. Decrease in abdominal pain (both at baseline and that associated with PO intake)

Secondary:

1. Decrease/elimination of pre-existing nausea/vomiting frequency and severity
2. Decrease/elimination of analgesic use
3. Background

   Experience with Procedure:

   CT-guided, celiac ganglion temporary block with liposomal bupivacaine. The PI, Dr. Georgiades has performed CT-guided nerve blocks hundreds of times, including celiac ganglion block, over the past 15 years. Nerve and specifically celiac ganglion block is an approved procedure for abdominal pain treatment, and is performed by Interventional Radiology at Johns Hopkins. Dr. Georgiades is a full time faculty in the Division of Interventional Radiology. He has privileges for performing CT-guided Celiac Ganglion block, as well as conscious sedation. Dr. Georgiades will be the only investigator performing this procedure in the test population.

   Clinical Data (with medication):

   Liposomal bupivacaine has long been used as an effective local analgesic, especially in orthopedic and plastic surgery.

   Clinical Data (Celiac ganglion block):

   Celiac ganglion block has been used for over a century for the treatment of abdominal pain. CT-guided celiac ganglion block has been introduced in the 1950s and most commonly performed with a combination of lidocaine and alcohol for permanent celiac ablation.

   Experience with Medication:

   Liposomal bupivacaine is an (food and drug administration) FDA approved drug and has long been used as a local anesthetic. It is simply a long acting formulation of bupivacaine. Bupivacaine's half-life is 2.7 hours. Since the procedure is performed under conscious sedation, the effects of bupivacaine cannot be distinguished from those of the medication given for sedation (Versed and fentanyl). The half-life of liposomal bupivacaine on the other hand, is approximately 24 hours. Therefore any symptom relief on post-test day #1 or 2 can be attributed to celiac ganglion blockade and not to sedation medication.

   Liposomal bupivacaine is available in 266 mg vials which is the maximum recommended single dose for adults.
4. Study Procedures a. Study design, including the sequence and timing of study procedures (distinguish research procedures from those that are part of routine care). The research protocol is highlighted in light brown below. All else is part of the patient's standard of care treatment. There are two potential patient populations than are candidates for the research protocol. 1. those with dysautonomia-related GI dysmotility, misdiagnosed as having MALS after MALS surgery fails to relieve symptoms, and 2. those with known dysautonomia-related dysmotility and related symptoms. The research procedure includes the CT-guided celiac ganglion block only. This test will be used to confirm (or exclude) dysautonomia as the patient's cause of GI symptoms. Those who have symptom relief after the test block, will proceed with open celiac ganglion resection.

Treatment Description:

1. SELECTION/RECRUITMENT

Potential Population Pool (PPP):

Adolescents and adults with diagnosis of :

1. Median Arcuate Ligament Syndrome (MALS)
2. Both MALS & Postural orthostatic Tachycardia Syndrome (POTS)
3. POTS or other Dysautonomia symptoms & bowel dysmotility

Study Population (Subgroup of PPP):

1. MALS patients with little or no improvement after laparoscopic arcuate ligament release
2. MALS & POTS patients with little or no improvement after laparoscopic arcuate ligament release
3. POTS/Dysautonomia patients with bowel dysmotility Symptoms: Required: Chronic nausea, food intolerance, abdominal pain, Additional: Chronic vomiting, need for enteral or parenteral Nutrition, hyperhidrosis, complex regional pain syndrome, Raynaud's Exclusion Criteria: Evidence for non-dysautonomia related causes of the patient's symptoms.

Must Exclude: Chronic cholecystitis, gastritis, peptic ulcer disease, gastro esophageal reflux, celiac disease, mesenteric atherosclerotic disease, vasculitis, anorexia, depression, other psych issues, etc Complete Compass 31 (Validated Autonomic Function Score)

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysautonomia-related GI dysmotility, misdiagnosed as having MALS after MALS surgery fails to relieve symptoms
* Patients with known dysautonomia-related dysmotility and related symptoms

Exclusion Criteria:

* Allergy to liposomal bupivacaine
* Platelets < 50 thousand
* International normalised ration (INR) > 1.7

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Amount of solid food intake by mouth per day | 2 days post celiac ganglion block
  Over the 2 days post Celiac Ganglion block, the investigators will monitor the patient (outpatient) for amount of solid food intake (grams) per day.
Change in abdominal pain as assessed by patient reported pain on scale 1-10 (10 worse) | Baseline and 2 days post-celiac ganglion block
  Patients with GI involvement of dysautonomia have abdominal pain which is worse with solid food intake. The patient's ability to take solid food without pain will be evaluated on scale 1-10 with 10 being worse pain.

SECONDARY OUTCOMES:
Number of episodes of nausea/vomiting per day | 2 days post celiac ganglion block
  The frequency of nausea/vomiting will be tabulated.
Change in amount of analgesic medications used | Baseline and 2 days post celiac ganglion block
  Patients with GI dysautonomia have chronic abdominal pain and take almost daily analgesic medication. The investigators shall evaluate the use of analgesic medication for the duration of the Celiac Ganglion block.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Georgiades, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No